CLINICAL TRIAL: NCT00914901
Title: Blood and Urinary Concentrations of Inhaled Salmeterol in Asthmatic Subjects and Elite Athletes With Asthma.
Brief Title: Concentrations of Salmeterol in Blood and Urine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Hormone Laboratory, Aker University Hospital, Oslo, Norway (Other)
Responsible Party: Jimmi Elers, Bispebjeg Hospital, Respiratory Research Unit
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SAL2009JE; EudraCT number 2009-012069-70
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Asthma
Keywords: Asthma; Doping; Salmeterol; Beta-agonist; Urine concentrations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy (Other): 10 healthy men
  Interventions: Drug: inhaled salmeterol
- Asthmatics (Other): 10 male asthmatic subjects
  Interventions: Drug: inhaled salmeterol
- Elite athletes with asthma (Other): 10 male elite athletes with asthma
  Interventions: Drug: inhaled salmeterol

INTERVENTIONS:
Drug: inhaled salmeterol — Inhalation of 100 micrograms salmeterol in one dose.

SUMMARY:
The purpose of the study is to assess the blood and urine concentrations of inhaled salmeterol.

DETAILED DESCRIPTION:
The purpose of the study is to assess the serum and urine concentrations of salmeterol after inhalation of 100 microgram salmeterol in one dose.

Furthermore, to evaluate any difference in three groups: 10 healthy men, 10 male asthmatic subjects and 10 male elite athletes with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma with positive reversibility or challenge test.
* Informed consent.
* Age between 18-45 years.
* Sex: male.
* Asthma classified as mild to moderate according to GINA guidelines.
* Used beta-2-agonist in minimum 12 months.

Exclusion Criteria:

* Smokers or ex-smokers with a smoking history of 10 pack years or more.
* Respiratory tract infections within the last 2 weeks prior to study day.
* Subjects with other chronic diseases than asthma and/or allergy.
* Allergy towards the study medicine.
* Use of beta-2-agonist 10 days prior to study day.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Serum and urine concentrations of salmeterol | baseline, 4, 8, and 12 hours after medicine administration

CONTACTS AND LOCATIONS:
Overall Officials: Jimmi Elers, MD, Principal Investigator — Bispebjerg Hospital, Respiratory Research Unit
Locations (1):
- Bispebjerg Hospital, Respiratory Research Unit, København NV, Denmark